CLINICAL TRIAL: NCT03056066
Title: Accuracy of Spircare Device as Compared to the Conventional Plethysmograph
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Spircare Ltd. (Industry)
Responsible Party: Sponsor
Other Study IDs: DA-1
Record Dates: First submitted 2017-02-13; First posted 2017-02-17 (Actual); Last update posted 2018-05-01 (Actual); Status verified 2018-04

CONDITIONS: COPD Asthma; Pulmonary Fibrosis
MeSH Terms: conditions — Pulmonary Fibrosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Plethysmograph — A full Body Plethysmography examination

SUMMARY:
The purpose of this study is to assess the accuracy of FRC and airway resistance calculate values of Spircare device as compared to the conventional body plethysmograph in healthy adults and patients with obstructive and restrictive pulmonary diseases/disorders.

ELIGIBILITY:
Inclusion Criteria:

1. Signed Informed consent.
2. Age≥18 year.
3. Subject is cooperative and capable of following instructions.
4. Phase I: Healthy asymptomatic subjects, never smokers without known history of respiratory, cardiovascular, hepatic, renal or metabolic disease.
5. Phase II: Chronic pulmonary patients with lung volume disorders:

   * COPD
   * Asthma
   * Restrictive diseases such as pulmonary fibrosis, other interstitial lung diseases, kyphoscoliosis, neuro-muscular disorders.

Exclusion Criteria:

1. Subjects unable or unwilling to give informed consent.
2. Subjects who are unable to satisfactorily perform routine, full lung function testing (due to non-compliance or claustrophobia).
3. History suggesting upper respiratory infection during the four weeks prior to testing
4. Physical activity during 1 hour prior to the Study.
5. Patients with a tracheostomy.
6. Pregnant women.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Phase I Health subjects without respiratory system disease.
  Phase II Subjects which are referred to a Pulmonary Functional Testing in the Meir pulmonary unit.
Sampling Method: Non-Probability Sample
Enrollment: 90 (Estimated)
Dates: Start 2017-07-31 (Actual); Primary Completion 2018-11 (Estimated); Study Completion 2019-01 (Estimated)

PRIMARY OUTCOMES:
The FRC and air way resistance values of the body plethysmograph will be compared to the values of the Spircare device | September 2017
  The primary outcome of the FRC and air way resistance of the Spircare device against the plethysmograph will be displayed as scatter plot. A linear regression and the R2 value will be display as well. The associated Bland-Altman plots comparing the FRC and airway resistance of the Spircare device to the plethysmograph with lines that represent width of 0.1 (±1.96*SD).

CONTACTS AND LOCATIONS:
Locations (1):
- "Meir" Medical Center, Kfar Saba, Israel

IPD SHARING:
Plan to Share IPD: Undecided